CLINICAL TRIAL: NCT00200369
Title: Characterization of the Adherence Threshold for HIV Suppression of a Kaletra-based Regimen
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Abbott (Industry)
Other Study IDs: 03-10-268; Abbott Laboratories #378-03-71
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infection
Keywords: HIV; Adherence; Antiretroviral therapy; Protease inhibitor; Lopinavir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: MEMS cap

SUMMARY:
The hypothesis of this study is that the level of adherence necessary to achieve HIV virologic suppression with a ritonavir boosted protease inhibitor regimen (i.e. lopinavir/ritonavir) is less than the 95% rate observed in the published literature with unboosted regimens.

DETAILED DESCRIPTION:
The existing dogma is that patients receiving highly active antiretroviral therapy (HAART) to treat their HIV infection must take at least 95% of prescribed doses in order to maintain full suppression of viral replication. This belief is largely based on a single study that was performed between 1997 and 1999 (Ann Int Med 2000;133:21-30). The vast majority of patients in this study were receiving regimens based on either indinavir, nelfinavir, ritonavir, or saquinavir. All of these agents have relatively short half-lives, and therefore must be taken on time two or three times per day. Newer medications such as lopinavir/ritonavir (Kaletra) feature much more favorable pharmacokinetic profiles. On the basis of improved pharmacokinetics, there is reason to believe that regimens built around such agents may be more forgiving of missed medication doses.

This study aims to enroll 90 patients from the MMC I.D. Clinic who are either receiving or are about to receive Kaletra. Patients who agree to participate will be furnished with a MEMS cap, a bottle cap that electronically records each time that the bottle is opened and stores the data for computer download, and will undergo electronic monitoring of their Kaletra adherence for a period of siz months. Adherence data will not be reviewed during the study, but at study end (and at interim time points), the investigators will analyze the MEMS cap data from patients who have completed the study in order to determine the threshold value of adherence necessary to achieve satisfactory rates (i.e. 70-80%) of complete virologic suppression.

An additional aim of the study is to collect specimens from patients receiving Kaletra based regimens who experience virologic failure and to archive them for possible studies of genotypic and phenotypic resistance in the future.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Receiving twice daily Kaletra at an FDA approved dosage
* Age>18 years
* CD4 and viral load available within seven day of enrollment
* Patient willingness to accept MEMS cap monitoring
* HIV genotype within 60 days of enrollment for patients with viral load>1000
* Patient willingness to grant informed consent and complete five study visits

Exclusion Criteria:

* Provider or patient deem it unlikely that Kaletra therapy will continue for the ensuing 24 weeks
* Prescription of any medication that is contraindicated for Kaletra recipients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Montefiore Medical Center Infectious Diseases Clinic with eligibility criteria as listed below.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2004-05; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center I.D. Clinic, The Bronx, New York, United States

REFERENCES:
- [Derived] Shuter J, Sarlo JA, Kanmaz TJ, Rode RA, Zingman BS. HIV-infected patients receiving lopinavir/ritonavir-based antiretroviral therapy achieve high rates of virologic suppression despite adherence rates less than 95%. J Acquir Immune Defic Syndr. 2007 May 1;45(1):4-8. doi: 10.1097/QAI.0b013e318050d8c2. PMID 17460469